CLINICAL TRIAL: NCT03712280
Title: A Randomized, Open-Label, Phase 2a Comparator Study to Assess the Pharmacodynamics, Safety and Pharmacokinetics of Oral Administration MNK6106 (L-Ornithine Phenylacetate) Versus Rifaximin in Subjects With Hepatic Cirrhosis and a History of Prior Episodes of Hepatic Encephalopathy
Brief Title: MNK6106 for Liver Disease (Hepatic Cirrhosis) That in the Past Has Affected the Brain (Hepatic Encephalopathy)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MNK61062107
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Hepatic Cirrhosis; Hepatic Encephalopathy (HE)
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy | interventions — Drug Evaluation; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A: MNK6106 2 grams (tid) (Experimental): Participants receive 2 tablets of MNK6106 three times daily (tid) for 5 days
  Interventions: Drug: MNK6106
- Group B: MNK6106 4 grams (bid) (Experimental): Participants receive 4 tablets of MNK6106 twice daily (bid) for 5 days
  Interventions: Drug: MNK6106
- Group C: MNK6106 4 grams (tid) (Experimental): Participants receive 4 tablets of MNK6106 tid for 5 days
  Interventions: Drug: MNK6106
- Group D: Rifaximin 550 mg (bid) (Active Comparator): Participants receive 1 tablet of rifaximin bid for 5 days
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: MNK6106 — 1 gram tablet of MNK6106 for oral administration
  Other Names: Study Drug; L-Ornithine Phenylacetate
  Arms: Group A: MNK6106 2 grams (tid); Group B: MNK6106 4 grams (bid); Group C: MNK6106 4 grams (tid)
Drug: Rifaximin — 550 mg tablet of rifaximin for oral administration
  Other Names: Xifaxan
  Arms: Group D: Rifaximin 550 mg (bid)

SUMMARY:
The main reason for this study is to see how the study drug interacts with the body.

It will compare different doses of the study drug with a drug already in use.

Participants will be adults with liver disease that has affected the brain in the past.

ELIGIBILITY:
Key Inclusion Criteria:

A potential participant may only be included if (at screening), he/she:

1. Understands the study and has signed informed consent
2. Is an adult, not pregnant or lactating
3. Has cirrhosis of the liver
4. Has had 1 instance of HE within 12 months
5. Has hyperammonaemia defined as ≥37 μmol/L at screening

Key Exclusion Criteria:

A potential participant will be excluded if (at screening), he/she:

1. Has contraindicated allergies
2. Expects liver transplant within 1 month
3. Has had a liver shunt within the last 3 months
4. Has inadequate kidney, gastrointestinal, or cardiac function
5. Has cancer, infection, lab abnormalities, or any other condition that, per protocol or in the opinion of the investigator might compromise:

   1. the safety and well-being of the participant or potential offspring
   2. the safety of study staff
   3. the analysis of results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (5):
- United States (4):
  - Southern California Research Center, Coronado, California
  - Inland Empire Clinical Trials, Rialto, California
  - Global Clinical Professionals, St. Petersburg, Florida
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
- Fundacion de Investigacion (Research Foundation), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03712280) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 50 participants were enrolled in the United States and Puerto Rico
Groups:
- Group A: MNK6106 2 Grams (Tid): Participants receive 2 (1 gm) tablets of MNK6106 three times daily (tid) for 5 days
- Group B: MNK6106 4 Grams (Bid): Participants receive 4 (1 gm) tablets of MNK6106 twice daily (bid) for 5 days
- Group C: MNK6106 4 Grams (Tid): Participants receive 4 (1 gm) tablets of MNK6106 tid for 5 days
- Group D: Rifaximin 550 mg (Bid): Participants receive 1 (500 mg) tablet of rifaximin bid for 5 days
Period: Overall Study
Arm/Group | Group A: MNK6106 2 Grams (Tid) | Group B: MNK6106 4 Grams (Bid) | Group C: MNK6106 4 Grams (Tid) | Group D: Rifaximin 550 mg (Bid)
Started (Participants randomized) | 12 | 12 | 13 | 13
Safety Population (All participants randomized and treated) | 12 | 11 | 13 | 12
Modified Intent to Treat Population | 12 | 11 | 13 | 12
Completed 5 Day Treatment | 11 | 11 | 12 | 12
Completed | 11 | 11 | 12 | 12
Not Completed | 1 | 1 | 1 | 1
Not completed — Randomized, but not treated due to Adverse Event | 0 | 1 | 0 | 1
Not completed — Withdrawal by Participant or Caregiver | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: MNK6106 2 Grams (Tid) | Group B: MNK6106 4 Grams (Bid) | Group C: MNK6106 4 Grams (Tid) | Group D: Rifaximin 550 mg (Bid) | Total
Number analyzed (Participants) | 12 | 11 | 13 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 10 | 11 | 42
  >=65 years | 1 | 1 | 3 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.10) | 58.2 (7.95) | 58.2 (10.56) | 55.2 (9.09) | 57.2 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 6 | 20
  Male | 6 | 8 | 8 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 7 | 10 | 35
  Not Hispanic or Latino | 1 | 4 | 6 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 10 | 11 | 11 | 11 | 43
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — All participants were enrolled in the United States and Puerto Rico. Puerto Rico was treated as part of the United States.
  participants
    United States | 12 | 11 | 13 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Ammonia Plasma Levels at Baseline and Day 5
Description: This test measures the level of ammonia in your blood. Ammonia, also known as NH3, is a waste product made by your body during the digestion of protein. Normally, ammonia is processed in the liver, where it is changed into another waste product called urea. Urea is passed from the body in urine.
  If your body cannot process or eliminate ammonia, a lab test of a blood sample shows it has built up in the bloodstream. High ammonia levels in the blood can lead to serious health problems, including hepatic encephalopathy.
Time Frame: Baseline, Day 5
Population: modified Intent to Treat (mITT)
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Group A: MNK6106 2 Grams (Tid) | Group B: MNK6106 4 Grams (Bid) | Group C: MNK6106 4 Grams (Tid) | Group D: Rifaximin 550 mg (Bid)
Number analyzed (Participants) | 12 | 11 | 13 | 12
μmol/L
  Baseline | 70.4 (23.4) | 91.4 (35.0) | 92.6 (34.7) | 78.1 (25.0)
  Day 5/Pre-Dose in the Morning: number analyzed (Participants) | 10 | 11 | 12 | 10
  Day 5/Pre-Dose in the Morning | 72.7 (21.8) | 63.9 (16.9) | 74.9 (21.9) | 75.8 (31.3)
  Day 5/4 Hours Post Morning Dose: number analyzed (Participants) | 11 | 11 | 10 | 10
  Day 5/4 Hours Post Morning Dose | 69.8 (27.7) | 60.9 (13.3) | 73.0 (11.5) | 71.6 (29.5)

2. Secondary Outcome: Number of Participants With Adverse Events by the End of the Trial
Description: End of trial is defined as 7 (+/-3) days after last study treatment
Time Frame: within 15 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: MNK6106 2 Grams (Tid) | Group B: MNK6106 4 Grams (Bid) | Group C: MNK6106 4 Grams (Tid) | Group D: Rifaximin 550 mg (Bid)
Number analyzed (Participants) | 12 | 11 | 13 | 12
Participants
  Affected by Serious Adverse Events | 0 | 0 | 2 | 0
  Affected by Any Non-serious Adverse Event | 5 | 6 | 9 | 5
  Affected by Non-serious Adverse Events in the 5% Reporting Threshold | 5 | 6 | 8 | 5

ADVERSE EVENTS:
Time Frame: within 15 days
Description: All serious adverse events are reported. Non-Serious Treatment-Emergent Adverse Events reported by 5% or more participants in any treatment group are reported.
Arm/Group | Group A: MNK6106 2 Grams (Tid) | Group B: MNK6106 4 Grams (Bid) | Group C: MNK6106 4 Grams (Tid) | Group D: Rifaximin 550 mg (Bid)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 2/13 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 6/11 | 8/13 | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: MNK6106 2 Grams (Tid) (N=12) | Group B: MNK6106 4 Grams (Bid) (N=11) | Group C: MNK6106 4 Grams (Tid) (N=13) | Group D: Rifaximin 550 mg (Bid) (N=12)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: MNK6106 2 Grams (Tid) (N=12) | Group B: MNK6106 4 Grams (Bid) (N=11) | Group C: MNK6106 4 Grams (Tid) (N=13) | Group D: Rifaximin 550 mg (Bid) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT03712280/Prot_SAP_000.pdf